CLINICAL TRIAL: NCT04887675
Title: A Single Centre, Prospective, Two-armed Magnetic Resonance Spectroscopy Study to Compare Imaging Biomarkers of Neuroinflammation and Neurodegeneration Between HIV-positive Subjects Switched and Initially Treated With INSTI
Brief Title: Neuroinflammation and Neurodegeneration in HIV-positive Subjects Switched and Initially Treated With INSTI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Novi Sad (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Snezana Brkic, Full Professor, Dean of Faculty of Medicine, University of Novi Sad
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UNoviSad
Record Dates: First submitted 2021-04-30; First posted 2021-05-14 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: HIV I Infection; HIV Associated Lipodystrophy; Metabolic Syndrome; Aging
MeSH Terms: conditions — HIV-Associated Lipodystrophy Syndrome; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients switched from PI/EFV based ART to INSTI based ART (Active Comparator): 60 patients on PI/EFV based ART, stable on treatment (undetectable viral load for at least 6 months). At the beginning of the study they are switched to INSTI based regimen. The reasons for the switch will be side effects or long-term toxicities like hyperlipidemia, diarrhea, (PI), insomnia, headache (EFV), high Framingham score (PI/EFV)
  Interventions: Diagnostic Test: MRI
- Patients initially treated with INSTI based regimens (Active Comparator): 60 patients initially started on INSTI based ART (raltegravir and dolutegravir), stable on treatment (undetectable viral load for at least 6 months).
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Both groups with undergo neuroimaging on 3T magnetic resonance unit (Trio Tim, Siemens, Erlangen, Germany) in the Center for Diagnostic Imaging, Oncology Institute of Vojvodina, Serbia. Multivoxel MRS will be performed in the supratentorial cerebral parenchyma, covering white matter of frontal and parietal lobes, as well as cortical grey matter in frontal and parietal lobes and the whole cingulate gyrus.

SUMMARY:
Since the HIV changed its course to the chronic disease, high incidence of metabolic syndrome both in HIV positive and negative subjects has become an issue. Given the successful peripheral suppression of HIV after introduction of combined antiretroviral therapy (cART), comorbidities associated with aging and cognitive functioning, play the main role in the overall quality of life and adherence to the therapy. Continuous low-level neuroinflammation results in continuous and diffuse neuronal death or dysfunction leading to a certain level of neurodegeneration. Additionally, metabolic syndrome contributes to neurodegeneration causing damage to the brain vasculature and provoking the ischemic incidents.

The aim of this study would be to explore the influence of switching to the INSTI based cART using neuroimaging biomarkers of inflammation and neurodegeneration. The second aim would be to monitor these neuroimaging biomarkers in patients receiving INSTI-based cART in a one-year follow-up period. Additionally, we would compare the markers of metabolic syndrome and cognitive functioning (executive functions) in HIV-positive patients after switching to INSTI-based cART and in HIV-positive patients receiving INSTI-based cART from the start.

This study represents a single-center, prospective, interventional, two-armed single study. Arm I will include 60 patients on PI/EFV based ART, stable on treatment, who are switched to INSTI based regimen at the beginning of the study due to side effects or long-term toxicities like hyperlipidemia, diarrhea, (PI), insomnia, headache (EFV), high Framingham score (PI/EFV). Arm II will include 60 patients initially on INSTI-based ART, stable on treatment. The same data sets will be collected for both groups of patients. The variables collected will be related to metabolic syndrome (levels of LDL and HDL cholesterol, triglycerides, fasting insulin, glucose, blood pressure, waist circumference, waist to hip and waist to height ratio), performance on neurocognitive tests and MR spectroscopy neuroinflammation and neurodegeneration markers at the beginning of the study, as well as in 12 months follow up. Presence of steatosis and visceral fat thickness will be assessed using ultrasonography of abdomen.

The primary imaging will be performed at the time of enrollment of patients, along with the neurocognitive testing and blood sampling. The secondary imaging (follow up) will be performed 12 months after the initial, also followed by neurocognitive assessment and blood sampling.

Anthropometric measurements will be acquired at the time of blood sampling. Statistical analysis will be performed after collecting the data. Our work could significantly contribute to the better life quality in the aging of HIV positive subjects in the domain of cognitive functioning, tightly associated with adherence and overall life quality.

DETAILED DESCRIPTION:
Serbia is low income country with epidemiology of HIV infection resembling those in developed countries, with average age of patients around 50 years and majority of them being the MSM population. Another important issue is the high incidence of metabolic syndrome both in HIV positive and negative subjects. With the successful peripheral suppression of HIV after introduction of combination antiretroviral therapy (cART), HIV disease has changed its course and now represents a chronic disease with majority of patients reaching senium. In these patients, comorbidities associated with aging, especially in the means of cognitive functioning, play the main role in the overall quality of life and adherence to the therapy. Considering the fact that viral particles of HIV remain latent in microglial cells and macrophages, virus only triggers the inflammatory response in the brain, which is afterwards maintained in the form of low-level neuroinflammation by the microglia and macrophages, resulting in continuous and diffuse neuronal death or dysfunction and leading to a certain level of neurodegeneration. With aging of HIV-positive subject, this form of neurodegeneration is combined with the physiological aging of the brain, most probably in the synergistic manner. Recent studies showed that this peripheral inflammation alters the blood-brain barrier and allows the penetration of HIV and particles, starting the "circulus vitiosus" all over again. Additionally, metabolic syndrome contributes to neurodegeneration causing damage to the brain vasculature and provoking the ischemic incidents.

The switch from the old fashion to the modern INSTI based cART and its influence on the process of neurodegeneration, as well as the role of neuroprotection of INSTI are still not well examined and documented. The aim of this study would be to explore the influence of switching to the INSTI based cART on neuroimaging biomarkers of inflammation and neurodegeneration obtained by MRS. The second aim would be to monitor these neuroimaging biomarkers in patients receiving INSTI based cART from the start in a one-year follow up period. Additionally, we would compare the markers of metabolic syndrome and cognitive functioning (executive functions) in HIV-positive patients after switching to INSTI based cART and in HIV-positive patients receiving INSTI based cART from the start.

This study represents a single-center, prospective, interventional, two-armed single study. Arm I will include 60 patients on PI/EFV based ART, stable on treatment, who will be switched to INSTI based regimen at the beginning of the study due to side effects or long-term toxicities like hyperlipidemia, diarrhea, (PI), insomnia, headache (EFV), high Framingham score (PI/EFV). Arm II will include 60 patients initially started on INSTI based ART, stable on treatment. The same data set will be collected in both groups of patients. The variables collected will be related to metabolic syndrome (levels of LDL and HDL cholesterol, triglycerides, fasting insulin, glucose, blood pressure, waist circumference, waist to hip and waist to height ratio), performance on neurocognitive tests and MRS neuroinflammation and neurodegeneration markers at the beginning of the study, as well as the 12 months after the beginning.

Besides the biochemical and anthropometric parameters of metabolic syndrome, presence of steatosis and visceral fat thickness will be assessed using ultrasonography of abdomen.

The primary imaging will be performed at the time of enrollment of patients. At the same time point, immediately before of after the imaging, patients will fulfill the neurocognitive testing. Blood samples will be taken within one week prior to imaging. The secondary imaging (follow up) will be performed 12 months after the initial, also followed by neurocognitive assessment in the same time relationship. Blood samples will be taken within one week prior to imaging.

Anthropometric measurements will be acquired at the time of blood sampling. Adequate statistical analysis will be performed after collecting the data. Our work could significantly contribute to the better life quality in the aging of HIV positive subjects in the domain of cognitive functioning, tightly associated with adherence and overall life quality.

ELIGIBILITY:
Inclusion Criteria:

* Male (in order to eliminate the hormonal influences on the levels of brain metabolites),
* older than 18 years,
* HIV seropositivity confirmed on PCR testing,
* undetectable viral load for over one year,
* conventional magnetic resonance imaging (MRI) normal.
* In group I, the additional criterion would be stable cART not containing INSTI for over one year.
* In group II, the inclusion criteria will be the INSTI base regimen introduced at least one year prior to imaging.

Exclusion Criteria:

* active infiltrative or infective/opportunistic neurological illness,
* chronic neurological diseases (multiple sclerosis, vascular and non-vascular dementia, other neurodegenerative conditions),
* active abuse of narcotic drugs,
* hepatitis B or C coinfection,
* deep white matter lesions (focal or diffuse, such as lacunar stroke, leukoaraiosis, infiltrative or infective foci, metastases etc.),
* International HIV Dementia Scale (IHDS) score <10 (only neuro-asymptomatic subjects would be included in the study), and
* contraindications for MRI examination

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Levels od inflammatory biomarkers in patients switched to INSTI based regimens | 1 year
  We will assess neuroimaging biomarkers obtained on magnetic resonance spectroscopy. These markers are: N-acetyl aspartate (NAA, marker of neuronal density and function), choline (Cho, marker of membrane metabolism and degradation), myoinositol (mI, marker of glial proliferation) and creatine (Cr, reference marker and marker of energy depot). These markers will be derived as ratios: NAA/Cr, Cho/Cr and mI/Cr.

SECONDARY OUTCOMES:
Performance performance on neurocognitive test in patients initially treated with INSTI based regimens | 1 year
  Neurocognitive testing will be performed using validated battery of neurocognitive tests (Montreal Cognitive Assessment, MoCA), consisted of relevant tests for memory deficits, executive functions, attention and concentration.
Incidence of metabolic syndrome in patients initially treated with INSTI based regimens | 1 year
  Metabolic syndrome incidence will be described using relevant statistical parameters (frequency and incidence rate).

CONTACTS AND LOCATIONS:
Overall Officials: Snezana Brkic, Principal Investigator — University of Novi Sad
Locations (1):
- Faculty of Medicine, University of Novi Sad, Novi Sad, Serbia

IPD SHARING:
Plan to Share IPD: No